CLINICAL TRIAL: NCT03929016
Title: A Phase I, Double-blind, Randomised, Single Centre, Parallel Group, Single-dose, Dose-escalation, Placebo Controlled Study of the Safety, Tolerability and Pharmacokinetics of DNDI-0690 After Oral Dosing in Healthy Subjects
Brief Title: Single Oral Dose Escalation Study of DNDI-0690 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DNDi-0690-01; 2018-002021-35 (EudraCT Number); QSC200932 (Other: Quotient Sciences)
Record Dates: First submitted 2019-04-09; First posted 2019-04-26 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Visceral Leishmaniasis; Cutaneous Leishmaniases
Keywords: First-in-human; single ascending dose; healthy volunteer
MeSH Terms: conditions — Leishmaniasis, Visceral; Leishmaniasis, Cutaneous

STUDY DESIGN:
Intervention Model Description: Single Ascending Dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Active DNDI-0690 male 10mg fasting (Experimental): Single dose 10mg male fasting
  Interventions: Drug: DNDI-0690
- Placebo male fasting (Placebo Comparator): Single dose placebo male fasting
  Interventions: Drug: Placebo of DNDI-0690
- Active DNDI-0690 male 30mg fasting (Experimental): Single dose 30mg male fasting
  Interventions: Drug: DNDI-0690
- Active DNDI-0690 male 150mg fasting (Experimental): Single dose 150mg male fasting
  Interventions: Drug: DNDI-0690
- Active DNDI-0690 male 400mg fasting (Experimental): Single dose 400mg male fasting
  Interventions: Drug: DNDI-0690
- Active DNDI-0690 male 1200mg fasting (Experimental): Single dose 1200mg male fasting
  Interventions: Drug: DNDI-0690
- Active DNDI-0690 male 3600mg fasting (Experimental): Single dose 3600mg male fasting
  Interventions: Drug: DNDI-0690
- Placebo male fed (Placebo Comparator): Placebo male fed
  Interventions: Drug: Placebo of DNDI-0690
- Active DNDI-0690 400mg male fed (Experimental): Single dose 400mg male fed
  Interventions: Drug: DNDI-0690
- Placebo female fasting (Placebo Comparator): Placebo female fasting
  Interventions: Drug: Placebo of DNDI-0690
- Active DNDI-0690 1200mg female fasting (Experimental): Single dose 1200mg female fasting
  Interventions: Drug: DNDI-0690

INTERVENTIONS:
Drug: DNDI-0690 — capsules of 10, 100 and 200 mg
  Arms: Active DNDI-0690 1200mg female fasting; Active DNDI-0690 400mg male fed; Active DNDI-0690 male 10mg fasting; Active DNDI-0690 male 1200mg fasting; Active DNDI-0690 male 150mg fasting; Active DNDI-0690 male 30mg fasting; Active DNDI-0690 male 3600mg fasting; Active DNDI-0690 male 400mg fasting
Drug: Placebo of DNDI-0690 — capsules of matching placebo
  Arms: Placebo female fasting; Placebo male fasting; Placebo male fed

SUMMARY:
This study will evaluate how the test medicine DNDI-0690 is taken up and broken down by the body and will also look at the safety and tolerability of the test medicine after a single dose. This is the first time the test medicine DNDI-0690 will be administered to humans.

DETAILED DESCRIPTION:
DNDI-0690 is intended to be used as oral treatment for Visceral Leishmaniasis with potential for the cutaneous form of the disease, Cutaneous Leishmaniasis. The present protocol describes the first-in-human (FIH) study with DNDI-0690.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males (Cohorts 1 to 7) or healthy WONCBP (Cohort 8)
* 18 to 55 years (Cohorts 1 to 7) or 18 to 60 years (Cohort 8)of age at the time of signing informed consent
* Body mass index (BMI) of 18.0 to 30.1 kg/m2 as measured at screening
* General good physical health determined by medical and surgical history, physical examination, 12-lead ECG, vital signs and clinical laboratory tests
* Normal blood pressure: Systolic blood pressure between ≥90 and ≤140 mmHg, Diastolic blood pressure ≤90 mmHg, measured after 10 min rest in supine position at screening, admission and pre-dose
* A resting Heart Rate (HR) between ≥40 and ≤90 bpm measured after 10 min rest in supine position at screening, admission and pre-dose
* ECG recording without clinically significant abnormality, including QTcF measure of ≤450 msec (male) or ≤470 msec (female) at screening, admission and pre-dose
* Having had no febrile seizures or infectious illness for at least 7 days prior to administration of the Investigational Medicinal Product (IMP)
* Must be willing and able to communicate and participate in the whole study
* Must provide written informed consent
* Must agree to adhere to the contraception requirements and life-style restrictions defined in the protocol

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the 3 months or 90 days prior to Day 1
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee
* Subjects who have previously been enrolled in this study and/or have received DNDI-0690 previously
* History of any drug or alcohol abuse in the past 2 years
* Demonstrating excess in caffeine/xanthine consumption (more than 6 cups of coffee or equivalent a day)
* Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type). As confirmed by a positive alcohol breath test at screening or admission
* Current smokers and those who have smoked within the last 12 months. As confirmed by a breath carbon monoxide reading of greater than 10 ppm at screening or admission
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
* Females of childbearing potential including those who are pregnant or lactating (all female subjects must have a negative serum pregnancy test at screening and admission). A woman is considered of childbearing potential unless she is permanently sterile (hysterectomy, bilateral salpingectomy, bilateral tubal ligation, bilateral tubal occlusion and bilateral oophorectomy) or is postmenopausal (had no menses for 12 months without an alternative medical cause and a serum follicle stimulating hormone [FSH] concentration ≥40 IU/L)
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening
* Clinically significant abnormal biochemistry, haematology, coagulation or urinalysis (especially aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transpeptidase (GGT), alkaline phosphatase (ALP), creatinine, and blood urea nitrogen (BUN)) as judged by the investigator (laboratory parameters are listed in Appendix 1). Subjects with Gilbert's syndrome are allowed
* Confirmed positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* Evidence of renal impairment at screening or admission, as indicated by an estimated creatinine clearance (CLcr) of <80 mL/min using the Cockcroft-Gault equation
* History of clinically significant cardiovascular, renal, hepatic, neurological (especially seizures), immunological, psychiatric, myopathies, bleeding tendency, respiratory and particularly gastrointestinal (GI) disease, especially peptic ulceration and chronic gastritis, GI bleeding, ulcerative colitis, Crohn's Disease or Irritable Bowel Syndrome, as judged by the investigator
* History of additional risk factors for Torsades des Pointe (eg heart failure, hypokalaemia, family history of long QT syndrome)
* Rare hereditary problems of fructose intolerance, glucose-galactose malabsorption or sucrose-isomaltase insufficiency
* Any relevant GI complaints within 7 days of dosing
* Subjects with a history of cholecystectomy or gall stones (Cohort 7 only)
* Serious adverse reaction or clinically relevant hypersensitivity to any drug or the formulation excipients (Hypromellose [HPMC], sodium lauryl sulphate [SLS], sucrose, croscarmellose sodium and magnesium stearate)
* Presence or history of clinically significant allergy requiring treatment (including asthma, urticaria, clinically significant allergic rash or other severe allergic diathesis), as judged by the investigator. Hay fever is allowed unless it is active
* Donation or loss of greater than 500 mL of blood within the previous 3 months or more than 100 mL within 30 days before signing Informed Consent Form (ICF) to this trial
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug (including anti-acid drugs) or vitamins/herbal remedies (eg St. John's Wort and others which are known to interfere with the Cytochrome P450 3A4 (CYP3A4) and P-glycoprotein (P-gp) metabolic pathways) or HRT in the 21 days before IMP administration. Administration of up to 4 g of paracetamol per day within 7 days of IMP administration is allowed
* Surgery within 12 weeks prior to screening, with the exception of appendectomy
* Any surgery (eg gastric bypass) or medical condition that may affect absorption of orally administered drugs
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of DNDI-0690 by Assessing the Occurrence of Treatment-emergent adverse events (TEAEs) | from baseline up to 7-10 days post-dose
  number of subjects experiencing TEAEs classified by MedDRA (Medical Dictionary for Regulatory Activities) System Organ Class and Preferred Terms
Safety and Tolerability of DNDI-0690 by Assessing the Changes in 12-lead electrocardiogram (ECG) parameters | from baseline up to 7-10 days post-dose
  corrected QT interval by Frideriecia's formula (QTcF) (msec)
Safety and Tolerability of DNDI-0690 by Assessing the Changes of Safety laboratory parameters related to liver function | from baseline up 7-10 days post-dose
  aspartate aminotransferase (AST)
Safety and Tolerability of DNDI-0690 by Assessing the Changes of Safety laboratory parameters related to liver function | from baseline up 7-10 days post-dose
  alanine aminotransferase (ALT)
Safety and Tolerability of DNDI-0690 by Assessing the Changes of Safety laboratory parameters related to renal function | from baseline up 7-10 days post-dose
  creatinine (mg/dL)
Safety and Tolerability of DNDI-0690 by Assessing the Changes of Safety laboratory parameters related to renal function | from baseline up 7-10 days post-dose
  creatinine clearance (CLcr)
Safety and Tolerability of DNDI-0690 by Assessing the Changes of Troponin I as a cardiac safety marker | 4h, 9h, 24h and 48h post-dose
  Troponin I

SECONDARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve (AUC) From Zero Extrapolated to Infinity (AUC0-inf) | pre-dose up to 72 hours post-dose
  To assess plasma pharmacokinetic parameters
Observed Maximum Concentration (Cmax) | pre-dose up to 72 hours post-dose
  To assess plasma pharmacokinetic parameters
Time to Maximum Observed Plasma Concentration (Tmax) | pre-dose up to 72 hours post-dose
  To assess plasma pharmacokinetic parameters
Apparent elimination half-life (T1/2) | pre-dose up to 72 hours post-dose
  To assess plasma pharmacokinetic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MD, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in the publication will be shared at the time of publication of study results.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: at the time of publication of study results.
Access Criteria: not yet defined